CLINICAL TRIAL: NCT05329961
Title: An Open-Label Clinical Trial Evaluating the Immunogenicity of the 9vHPV Vaccination 2-dose Regimen Over a Four-year Follow up Among Children 4 to 8 Years Old, An Exploratory Immunogenicity Study
Brief Title: Immunogenicity of the 9vHPV Vaccination 2-dose Regimen Among Children 4 to 8 Years Old
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Eilsha Wachman, Professor of Pediatrics, Vice Chair for Research, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-41686
Record Dates: First submitted 2022-03-21; First posted 2022-04-15 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Human Papilloma Virus
Keywords: Gardasil 9; Immunogenicity; Children
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): HPV 9-valent human papillomavirus vaccine (Gardasil 9) - 0.5mL intramuscular dose - 2 doses (Month 0, 12)
  Interventions: Drug: Gardasil9

INTERVENTIONS:
Drug: Gardasil9 — The Gardasil 9 vaccine is a recombinant L 1 VLP vaccine containing HPV types 6, 11,16,18, 31, 33, 45, 52 and 58 VLP. The vaccine is not currently licensed for children under 9 years of age but it is licensed in the USA for males and females ages 9 to 45 years old.
  Other Names: GARDASIL®

SUMMARY:
This study is an open-label nonrandomized exploratory proof of concept and descriptive 4-year immunogenicity study to assess immunogenicity after administration of a 2-dose regimen of 9-valent human papillomavirus vaccine (9vHPV) vaccine separated by 12 months (months 0, 12).

DETAILED DESCRIPTION:
Study participants will include 150 boys and girls aged 4-8 years (total, 75 boys and 75 girls) to receive 2 doses of the 9vHPV vaccine at 0 and 12 months. Patients will be recruited by age-group to achieve balanced enrollment of 15 girls and 15 boys per year of age. The investigators will examine the immunogenicity profile in this cohort, for which titers will be analyzed one month after dose 2 (Month 13) and at Month 60.

Though clinical efficacy cannot be assessed in young children because of limited exposure to human papillomavirus (HPV), this descriptive study will allow the investigators to understand whether the 9vHPV vaccine in younger patients provides immunogenicity similar to that shown for the 9-14 and 16-26 age groups who have received the 9vHPV vaccine.13 This study will require an IND for the use of the HPV vaccine in children younger than 9 years.

Immunogenicity will be measured by examining serum antibodies of all participants using a competitive Luminex immunoassay (cLIA).15 Month 60 serology will be by cLIA and IgG LIA assays. The antibody response testing will be performed at Merck Research Laboratory.

The goal of this study is to explore whether a 2-dose 9vHPV vaccine regimen with dosage separated by 12 months is immunogenic among children aged 4-8 years. The primary outcome will be geometric mean titers (GMT) for HPV6, HPV11, HPV16, HPV18, HPV31, HPV33, HPV45, HPV52, and HPV58 antibodies at months 13 and 60. Results will allow the investigators to qualitatively compare immunogenicity in individuals vaccinated at age 4-8 years to known immunogenicity in 9vHPV recipients vaccinated at ages 9-14.13 Knowledge of whether vaccination in this age group is sufficient to induce high-level protective antibody titers through 4 years after the second dose will support further efficacy studies in a larger randomized trial of a 2-dose 9vHPV regimen for children aged 4-8 years.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-8 years old
2. Receives care at the Boston Medical Center or one of the affiliated Community heath centers
3. Naïve to HPV Vaccine

Exclusion Criteria:

1. A history of severe allergic reaction, including known allergy to any vaccine component, specially severe allergic reaction to yeast
2. Immunocompromised/previous immunosuppressive therapy
3. Thrombocytopenia or other coagulation disorder

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
HPV6 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV6 if it is >30mMu.
HPV11 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV11 if it is >16mMu.
HPV16 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV16 if it is >20mMu.
HPV18 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV18 if it is >24 mMU.
HPV31 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV31 if it is >10 mMU.
HPV33 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV33 if it is >8 mMU.
HPV45 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV45 if it is >8 mMU.
HPV52 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV52 if it is >8 mMU.
HPV58 antibodies at 13 months | 13 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV58 if it is >8 mMU.
HPV6 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV6 if it is >30mMU.
HPV11 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV11 if it is >16 mMU.
HPV16 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV16 if it is >20 mMU.
HPV18 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV18 if it is >24mMU.
HPV31 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV31 if it is >10 mMU.
HPV33 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV33 if it is >8 mMU.
HPV45 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV45 if it is >8 mMU.
HPV52 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV52 if it is >8 mMU.
HPV58 antibodies at 60 months | 60 months
  A serum sample will be analyzed using 9-valent Luminex immunoassay (cLIA, mMU/mL) to assess the geometric mean for HPV antibodies. The results will be considered positive for HPV58 if it is >8 mMU.

SECONDARY OUTCOMES:
Injection site swelling after first injection | day 3 after injection
  Solicited local swelling will be graded from 0-4 where 0 is no swelling and 4 is severe swelling.
Injection site swelling after second injection | day 3 after injection
  Solicited local swelling will be graded from 0-4 where 0 is no swelling and 4 is severe swelling.
Injection site redness after first injection | day 3 after injection
  Solicited local redness will be graded from 0-4 where 0 is no redness and 4 is severe redness.
Injection site redness after second injection | day 3 after injection
  Solicited local redness will be graded from 0-4 where 0 is no redness and 4 is severe redness.

CONTACTS AND LOCATIONS:
Overall Officials: Elisha Wachman, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No